CLINICAL TRIAL: NCT05298891
Title: Deciphering the Role of a Low Protein Diet in Disease Control in Acromegalic Patients
Brief Title: Hypoproteic Diet in Acromegaly
Acronym: IpoProAcro
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Associated Prof. in Clinical Nutrition and MD, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 008/22
Record Dates: First submitted 2022-03-18; First posted 2022-03-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acromegalic adult in therapy with somatostatin analogues (Experimental): Patients will continue the usual medical outpatient visits cadency and will keep the same pharmacological therapy throughout the whole duration of the study. Drugs have to include somatostatin analogues. At the same time, patients will be trained by an expert dietician in the habit of an isocaloric and hypoproteic diet and will come back at 2,4,6 and 8 weeks after T0 for all the necessary study assessments and compliance checking.
  Interventions: Other: Usual clinical practice + hypoproteic diet

INTERVENTIONS:
Other: Usual clinical practice + hypoproteic diet — Diet will be composed by:
  * energy equal to daily energy expenditure (estimated by indirect calorimetry * physical activity factor)
  * fats 28-35%
  * carbohydrates 50-60%
  * proteins 0,7-0,8g/kg of body weight 10-13% Diet will be given to the patient after the first visit and the study will start once the patient begins the diet.

SUMMARY:
Since protein and AAs are master regulator of GH and IGF-I secretion, we hypothesized that a low protein diet could reduce GH and IGF-I levels in acromegalic patients in addition to conventional therapy. Furthermore, we aim to explore metabolomic, microbiota, and micro-vesicle fingerprints of GH hypersecretion during conventional therapy and after a low protein diet

DETAILED DESCRIPTION:
Nutrients are crucial modifiers of the GH/IGF-I axis. In particular, a close cross-talk between proteins and amino acids (AAs) and GH/IGF-I secretion exists.

Both AAs and proteins affect GH secretion. AAs stimulate GH secretion upon oral administration, with different potency among studies, being the combination of arginine and lysine the most powerful. Soy proteins also stimulate GH secretion when ingested either as hydrolysed proteins or free AAs. Furthermore, the acute GH response to AAs ingestion may be influenced by the daily amount of dietary protein/AAs consumption: diets high in proteins apparently increase basal GH levels.

AAs and proteins have a positive effect on IGF-I secretion as well. In general, high levels of proteins, especially animal and dairy proteins, and consumption of branched chain amino acids (BCAAs) increase serum IGF-I levels.

Considering pathological GH conditions, metabolomic analysis of acromegalic patients suggests that the main metabolic fingerprint of GH hypersecretion is a reduction in BCAAs, related to the disease activity. Moreover, there is evidence that GH, rather than IGF-I, is the main mediator of such metabolic fingerprint, which may be related to increased uptake of BCAAs by the muscles, increased gluconeogenesis, and raised consumption of BCAAs.

Thus, in acromegaly, a tailored diet is a further strategy that may contribute to blunt GH/IGF-I secretion. Indeed, some authors recently suggested that "personalized" or "precision" nutrition in some conditions and diseases could have an impact on their phenotype, combining dietary recommendations with individual's genetic makeup, metabolic and microbiome characteristics, and environment. However, studies on precision nutrition in acromegaly are still in a neonatal era.

ELIGIBILITY:
Inclusion Criteria:

* Age 18/65
* Diagnosis of Acromegaly
* In therapy with somatostatin analogues

Exclusion Criteria:

* pregnancy or lactation
* alchool or drugs abuse
* cancer
* Hematological diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in disease related hormones | Change from Baseline GH, IGF-1, IGFBP1, IGFBP3 blood levels at 15 days, 30 days, 45 days, 60 days
  Variation of GH, IGF-1, IGFBP1, IGFBP3 hormones

SECONDARY OUTCOMES:
Change in weight | Change from Baseline BMI at 15 days, 30 days, 45 days, 60 days
  Variation of body weight assessed through body mass index change (BMI)(kg/m2)
Change in body circumferences | Change from Baseline circumferences at 15 days, 30 days, 45 dyas, 60 days
  Variation of body circumferences (waist, hips)
Change in metabolic control | Change from Baseline lipid profile at 15 days, 30 days, 45 days, 60 days
  Change of cardio-metabolic risk factors: lipid profile
Change in metabolic control | Change from Baseline lipid profile at 60 days
  Change of cardio-metabolic risk factors: insulin resistance (HOMA-IR)
Change in kidney profile | Change from Baseline Serum Creatinin at 15 days, 30 days, 45 days, 60 days
  Variation of serum creatinin
Change in liver profile | Change from Baseline Serum Creatinin at 15 days, 30 days, 45 days, 60 days
  Variation of liver markers(AST, ALT, GGT)
Change in uric acid | Change from Baseline uric acid in blood at 15 days, 30 days, 45 days, 60 days
  Variation of uric acid in blood through enzymatic determination
Change in body composition | Change from Baseline fat mass% at 60 days
  Change of body composition (fat mass %) (BIVA)
Change in body composition | Change from Baseline fat mass% at 60 days
  Change of body composition (fat mass %) (DXA)
Change in blood count | Change from Baseline blood count at 15 days, 30 days, 45 days, 60 days
  Variation of blood count
Change in microbiota | Change from Baseline of prevalence of microbiota phyla at 15, 30 days, 45 days, 60 days
  Variation of prevalence of microbiota phyla through DNA sequencing of stools
Change in omics profile | Change from Baseline omic profile of stools at 15, 30 days, 45 days, 60 days
  Variation of lipidomic profile of stools through liquid and gas chromatography
Change in omics profile | Change from Baseline omic profile of stools at 15, 30 days, 45 days, 60 days
  Variation of proteomic profile of stools through liquid and gas chromatography
Change in microvesicles | Change from Baseline microvesicles levels at 15, 30 days, 45 days, 60 days
  Variation of urinary microvesicles levels
Change in microvesicles | Change from Baseline microvesicles levels s at 15, 30 days, 45 days, 60 days
  Variation of serum microvesicles levels
Change in basal metabolic rate | Change from Baseline basal metabolic rate at 60 days
  Variation of basal metabolic rate (kcal)

CONTACTS AND LOCATIONS:
Locations (1):
- : Italy Pediatric Endocrine Service of AOU Maggiore della Carità of Novara; SCDU of Pediatrics, Department of Health Sciences, University of Eastern Piedmont, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Caputo M, Pigni S, Agosti E, Daffara T, Ferrero A, Filigheddu N, Prodam F. Regulation of GH and GH Signaling by Nutrients. Cells. 2021 Jun 2;10(6):1376. doi: 10.3390/cells10061376. PMID 34199514
- [Background] Suminski RR, Robertson RJ, Goss FL, Arslanian S, Kang J, DaSilva S, Utter AC, Metz KF. Acute effect of amino acid ingestion and resistance exercise on plasma growth hormone concentration in young men. Int J Sport Nutr. 1997 Mar;7(1):48-60. doi: 10.1123/ijsn.7.1.48. PMID 9063764
- [Background] van Vught AJ, Nieuwenhuizen AG, Brummer RJ, Westerterp-Plantenga MS. Effects of oral ingestion of amino acids and proteins on the somatotropic axis. J Clin Endocrinol Metab. 2008 Feb;93(2):584-90. doi: 10.1210/jc.2007-1784. Epub 2007 Nov 20. PMID 18029456
- [Background] Sellini M, Fierro A, Marchesi L, Manzo G, Giovannini C. [Behavior of basal values and circadian rhythm of ACTH, cortisol, PRL and GH in a high-protein diet]. Boll Soc Ital Biol Sper. 1981 May 15;57(9):963-9. Italian. PMID 6269563
- [Background] Levine ME, Suarez JA, Brandhorst S, Balasubramanian P, Cheng CW, Madia F, Fontana L, Mirisola MG, Guevara-Aguirre J, Wan J, Passarino G, Kennedy BK, Wei M, Cohen P, Crimmins EM, Longo VD. Low protein intake is associated with a major reduction in IGF-1, cancer, and overall mortality in the 65 and younger but not older population. Cell Metab. 2014 Mar 4;19(3):407-17. doi: 10.1016/j.cmet.2014.02.006. PMID 24606898
- [Background] Allen NE, Appleby PN, Davey GK, Kaaks R, Rinaldi S, Key TJ. The associations of diet with serum insulin-like growth factor I and its main binding proteins in 292 women meat-eaters, vegetarians, and vegans. Cancer Epidemiol Biomarkers Prev. 2002 Nov;11(11):1441-8. PMID 12433724
- [Background] Hoppe C, Udam TR, Lauritzen L, Molgaard C, Juul A, Michaelsen KF. Animal protein intake, serum insulin-like growth factor I, and growth in healthy 2.5-y-old Danish children. Am J Clin Nutr. 2004 Aug;80(2):447-52. doi: 10.1093/ajcn/80.2.447. PMID 15277169
- [Background] Romo Ventura E, Konigorski S, Rohrmann S, Schneider H, Stalla GK, Pischon T, Linseisen J, Nimptsch K. Association of dietary intake of milk and dairy products with blood concentrations of insulin-like growth factor 1 (IGF-1) in Bavarian adults. Eur J Nutr. 2020 Jun;59(4):1413-1420. doi: 10.1007/s00394-019-01994-7. Epub 2019 May 14. PMID 31089868
- [Background] Beasley JM, Gunter MJ, LaCroix AZ, Prentice RL, Neuhouser ML, Tinker LF, Vitolins MZ, Strickler HD. Associations of serum insulin-like growth factor-I and insulin-like growth factor-binding protein 3 levels with biomarker-calibrated protein, dairy product and milk intake in the Women's Health Initiative. Br J Nutr. 2014 Mar 14;111(5):847-53. doi: 10.1017/S000711451300319X. Epub 2013 Oct 7. PMID 24094144
- [Background] Li R, Ferreira MP, Cooke MB, La Bounty P, Campbell B, Greenwood M, Willoughby DS, Kreider RB. Co-ingestion of carbohydrate with branched-chain amino acids or L-leucine does not preferentially increase serum IGF-1 and expression of myogenic-related genes in response to a single bout of resistance exercise. Amino Acids. 2015 Jun;47(6):1203-13. doi: 10.1007/s00726-015-1947-8. Epub 2015 Mar 5. PMID 25740607
- [Background] Coopmans EC, Berk KAC, El-Sayed N, Neggers SJCMM, van der Lely AJ. Eucaloric Very-Low-Carbohydrate Ketogenic Diet in Acromegaly Treatment. N Engl J Med. 2020 May 28;382(22):2161-2162. doi: 10.1056/NEJMc1915808. No abstract available. PMID 32459928